CLINICAL TRIAL: NCT01480609
Title: An Open Label, Single-dose, Fixed Sequence, Two Treatment Period Study to Assess the Effect of Haemodialysis on the Pharmacokinetics of Ezogabine/Retigabine and the N-acetyl Metabolite of Ezogabine/Retigabine (NAMR).
Brief Title: Effect of Haemodialysis on the Pharmacokinetics of Ezogabine/Retigabine and Its N-acetyl Metabolite
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115214
Record Dates: First submitted 2011-10-27; First posted 2011-11-29 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose-Dialysis (Active Comparator): Subjects will be dosed with study drug followed by a scheduled dialysis session
  Interventions: Drug: Retigabine / Ezogabine
- Dialysis-Dose (Active Comparator): Subjects will be dosed following the completion of their scheduled dialysis session
  Interventions: Drug: Retigabine / Ezogabine

INTERVENTIONS:
Drug: Retigabine / Ezogabine — Retigabine / Ezogabine will be available as immediate release tablets of 50 milligrams strength. Subjects will be administered the tablet will 250 milliliters of water

SUMMARY:
This in an open-label, single dose, fixed sequence, two treatment period study enrolling 8 patients (to obtain 6 evaluable) with end stage renal disease (ESRD) receiving haemodialysis. Patients will remain in the unit during each treatment period from admission to the collection of the final PK sample. The doses of ezogabine/retigabine in the two treatment periods will be separated by at least 7 days.

DETAILED DESCRIPTION:
Treatment Period 1: Subjects will be admitted on Day -1 when baseline assessments will be performed. On Day 1 subjects will receive a single dose of 100mg ezogabine/retigabine immediate release (IR) and dialysis will start 4 hours post-dose. Pharmacokinetic (PK) samples will be collected up to approximately 68 hours post-dose.

Samples of dialysate will be collected in 0-1, 1-2, 2-3, and 3-4 hour (if available) aliquots, timed from the start of dialysis. The volume of dialysate collected in each aliquot will be recorded.

Four samples of predialyzer ("arterial" line) blood and four samples of postdialyzer ("venous" line) blood will be obtained during the haemodialysis procedure at approximately one hour intervals starting immediately prior to the start of the procedure and finishing at the end of the procedure.

Subjects will be discharged from the unit following the collection of the last PK sample.

Treatment Period 2: Subjects will be admitted on Day -1 when baseline assessments will be performed. On Day 1 following the completion of their scheduled dialysis session subjects will receive a single dose of 100mg ezogabine/retigabine IR. PK samples will be collected up to approximately 68 hours post-dose.

Subjects will be discharged from the unit following the collection of the last PK sample.

In both treatment periods, PK blood samples will be obtained pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60 and 68 hours (or just prior next dialysis session - whichever is sooner) post-dose. Subjects will be discharged after the final post-dose draw.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older, at the time of signing the informed consent.
* ESRD patients with minimal or no residual renal function and receiving stabilised haemodialysis regimen.
* Body mass index with the range of 18-42 kg/m2 at screening.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods listed.
  * Child-bearing potential and agrees to use one of the contraception methods listed. Female subjects must agree to use contraception until at least 1 week post-last dose.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed. This criterion must be followed from the time of the first dose of study medication until at least 1 week post-last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Subjects with fluctuating or rapidly deteriorating condition that is not adequately controlled by medications
* Subjects with signs of a clinically significant infection.
* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months. Has history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt.
* Subjects with any other medical condition which, in the judgement of the investigator and medical monitor, could jeopardize the integrity of the data derived from that subject or the safety of the subject
* Clinically relevant laboratory or physical examination abnormalities (except for renal function tests or deviation of clinical laboratory values that are related to renal impairment).
* Subjects with blood pressure, after resting for ≥ 3 minutes, higher than 160/95 mmHg or lower than 100/50 mmHg. The patients receiving anthihypertensive treatment need to be on a stabilised treatment for three months.
* The screening ECGs measurements must be within the limit indicated in the protocol.
* Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.
* History of hemoglobinopathy.
* A radiological test involving contrast dye within 4 weeks prior to screening.
* Poor peripheral venous access.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Pregnant females
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2012-04-24 (Actual); Study Completion 2012-04-24 (Actual)

PRIMARY OUTCOMES:
Clearance (Cl/F), clearance during dialysis (CLD) and fraction of total clearance attributed to dialysis (FD) of ezogabine/retigabine and NAMR | During Dialysis (0-1, 1-2, 2-3, and 3-4 hour)
  Pharmacokinetic parameters
AUC(0-t), AUC (0-∞), T½, Cmax, Tmax of ezogabine/retigabine and NAMR in plasma. Amount of ezogabine/retigabine and NAMR cleared by dialysis (AD) | 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60 and 68 hours
  Pharmacokinetic parameters

SECONDARY OUTCOMES:
Nmber of Safety and tolerability parameters, including adverse event, clinical laboratory, and vital signs assessments | Participants will be assessed for the duration of the study - an expected average of 3 weeks
  Safety Parameters

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115214 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115214?search=study&search_terms=115214#rs
- Available data/document: Informed Consent Form: 115214 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115214 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115214 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115214 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115214 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115214 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115214 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register